CLINICAL TRIAL: NCT02764749
Title: Sustained Effects of Cranberry (Poly)Phenol Consumption on Vascular Function in Healthy Individuals
Brief Title: Cranberry (Poly)Phenol Consumption on Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Investigator of Division of Cardiology, Pulmonary Diseases, Vascular Medicine, Heinrich-Heine University, Duesseldorf
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Cranberry; 15-042 (Other: CTSU)
Record Dates: First submitted 2016-05-04; First posted 2016-05-06 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Young
Keywords: vascular function; endothelial function; polyphenols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- freeze dried powder whole cranberry dissolved in water (Experimental): Dietary Supplement: freeze dried cranberry powder
  Interventions: Dietary Supplement: cranberry (poly)phenol containing supplement
- freeze dried cranberry deprived powder dissolved in water (Placebo Comparator): Placebo comparator: freeze dried cranberry deprived powder
  Interventions: Dietary Supplement: Placebo comparator: cranberry (poly)phenol deprived supplement

INTERVENTIONS:
Dietary Supplement: cranberry (poly)phenol containing supplement — Sustained intake of 9 grams of freeze-dried cranberry powder per day (2x 4.5 grams daily over 1 month). The powder is dissolved in water and administered as a drink.
  Arms: freeze dried powder whole cranberry dissolved in water
Dietary Supplement: Placebo comparator: cranberry (poly)phenol deprived supplement — Sustained intake (2x 4.5 grams daily over 1 month) of a control supplement dissolved in water
  Arms: freeze dried cranberry deprived powder dissolved in water

SUMMARY:
Epidemiological studies suggest that the consumption of (poly)phenols rich foods such as cocoa, tea, fruits and vegetables is associated with lower blood pressure, reduced cholesterol and decreased cardiovascular risk. Cranberries are a rich source of (poly)phenols, including anthocyanins, proanthocyanidins and phenolic acids. Whether cranberries can improve vascular function when given over relevant time periods and in relevant populations is not known. Therefore, it is the overall hypothesis of the study proposal that chronic consumption of cranberries can improve endothelial function, a prognostically validated surrogate of cardiovascular risk. This study also aims to reveal which cranberry (poly)phenols have bioactive properties in healthy men. Consequently, plasma and urine metabolite peaks will be correlated with vascular outcomes and genome-wide expression microarrays will be performed to reveal cell signaling pathways associated with cranberry (poly)phenol-mediated cardioprotective events.

ELIGIBILITY:
Inclusion Criteria:

* healthy male subjects (no clinical signs or symptoms of CVD)
* Young >18 years, <35 years

Exclusion Criteria:

* CVD
* acute inflammation
* cardiac arrhythmia
* renal failure
* heart failure (NYHA II-IV)
* diabetes mellitus
* CRP > 1 mg/dl
* malignant disease

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change form Baseline Endothelial function at 1 month | 2 hours and 1 month
  Measured by Flow mediated dilation (FMD)

SECONDARY OUTCOMES:
Pulse wave velocity | Baseline and 1 month
  Measured by SphygmoCor 0 and 2 hours postconsumption
Blood pressure | Baseline and 1month
  automatical measurements 0 and 2 hours postconsumption
high density lipoproteins (HDL) | Baseline and 1 month
  measured on baseline and after 1 month
low density lipoproteins (LDL) | Baseline and 1 month
  measured on baseline and after 1 month
triglyceride | Baseline and 1 month
  measured on baseline and after 1 month

OTHER OUTCOMES:
Plasma cranberry (poly)phenol metabolites | Baseline and 1 month
  Measured by liquid chromotography- mass spectrometry (LC/MS) 0 and 2 hours postconsumption
Urinary cranberry (poly)phenol metabolites | Baseline and 1 month
  Measured by liquid chromotography- mass spectrometry (LC/MS) 0 and 2 hours postconsumption

CONTACTS AND LOCATIONS:
Overall Officials: Ana Rodriguez-Mateo, PhD, Principal Investigator — Division of Cardiology, Pulmonology and Vascular Medicine, University Hospital Duesseldorf
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, University Hospital Duesseldorf, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heiss C, Istas G, Feliciano RP, Weber T, Wang B, Favari C, Mena P, Del Rio D, Rodriguez-Mateos A. Daily consumption of cranberry improves endothelial function in healthy adults: a double blind randomized controlled trial. Food Funct. 2022 Apr 4;13(7):3812-3824. doi: 10.1039/d2fo00080f. PMID 35322843
- [Derived] Mena P, Favari C, Acharjee A, Chernbumroong S, Bresciani L, Curti C, Brighenti F, Heiss C, Rodriguez-Mateos A, Del Rio D. Metabotypes of flavan-3-ol colonic metabolites after cranberry intake: elucidation and statistical approaches. Eur J Nutr. 2022 Apr;61(3):1299-1317. doi: 10.1007/s00394-021-02692-z. Epub 2021 Nov 9. PMID 34750642